CLINICAL TRIAL: NCT02603939
Title: Understanding Pain Perception in Osteoarthritis: a Mechanistic Study in People With Knee Osteoarthritis
Brief Title: Understanding Pain Perception in Osteoarthritis
Acronym: PAPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 12.0056
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis; Pain
Keywords: Pain; Magnetic resonance imaging
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collected
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants with Advanced Knee OA: People with advanced knee osteoarthritis requiring joint replacement surgery are being assessed for their pain responses before and after joint replacement surgery
  Interventions: Procedure: Joint replacement surgery
- Participants with Early Knee OA: Participants with osteoarthritis with early disease who do not require joint replacement surgery are being assessed for pain

INTERVENTIONS:
Procedure: Joint replacement surgery — We are assessing pain responses in participants with osteoarthritis before an after joint replacement surgery
  Groups: Participants with Advanced Knee OA

SUMMARY:
Osteoarthritis (OA)is a painful and disabling disease, predicted to be the fourth largest cause of disability worldwide by 2020. It commonly affects the hip or knee ultimately resulting in total joint replacement. In order to assess disease progression and plan surgery, x-rays are taken as part of routine practice. However x-rays provide limited information about formation of substructures and changes occurring during progression of disease. The proposed study aims to invite patients with OA of the hip or knee to participate in detailed examinations of their pain and their painful joint through interviews, blood and urine samples taken, MRI magnetic resonance imaging)and donating their waste tissue after joint surgery (all of old joint). Informed patient consent will be sought in all cases.

DETAILED DESCRIPTION:
The patient will be asked for permission for a clinician to access their notes for information relevant to the research, including full medical history, their sex and date of birth. Tissue obtained from joint replacement surgery at St. George's Hospital and transferred to St.George's, University of London where it will be prepared for various experiments including looking at the genes and proteins in people with osteoarthritis. The blood and urine samples will also be taken to St. George's, University of London, and prepared for studies on the genes and proteins in people with osteoarthritis. All samples provided will be anonymised with no patient details on the samples and stored in locked freezers, in locked labs. at St.George's, University of London.

ELIGIBILITY:
Inclusion criteria:

Inclusion Criteria for OA patients:

Study participant will be recruited from rheumatology outpatient clinics and primary care:

1. fulfilling the American College of Rheumatology (ACR) criteria for the diagnosis of knee osteoarthritis
2. male or female,
3. symptomatic knee pain
4. on usual care for knee osteoarthritis including paracetamol and/or non-steroidal anti-inflammatory drugs
5. participants between 35 and 90 who will be undergoing knee replacement surgery or arthroscopy for osteoarthritis or knee surgery for fractured tibia/femur/fibula with osteoarthritis

Inclusion criteria for Early OA Patients

Study participant will be recruited from rheumatology outpatient clinics and primary care:

1. fulfilling the American College of Rheumatology (ACR) criteria for the diagnosis of knee osteoarthritis
2. male or female,
3. symptomatic knee pain
4. on usual care for knee osteoarthritis including paracetamol and/or non-steroidal anti-inflammatory drugs
5. Participants between 35 and 90 who have osteoarthritis but will not be undergoing knee surgery

Inclusion criteria for Healthy control subjects

1. Participants aged between 35 and 90 who do not have knee pain or osteoarthritis as a comparator group

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with symptomatic knee osteoarthritis who are in pain and are being considered for joint replacement surgery
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain outcomes measured by Western Ontario and McMaster Universities Index (WOMAC) | 1 Year after joint replacement
  Western Ontario and McMaster Universities Index (WOMAC)

SECONDARY OUTCOMES:
Magnetic Resonance Imaging Knee Osteoarthritis Score | Pre-operatively
  Level of tissue damage quantified by MOAKS scoring at baseline before joint surgery

CONTACTS AND LOCATIONS:
Overall Officials: Nidhi Sofat, MBBS, PhD, Principal Investigator — St George's, University of London
Locations (1):
- Hotung Centre for Musculoskeletal Diseases, London, United Kingdom